CLINICAL TRIAL: NCT01913730
Title: A PHASE II MULTI-CENTRE, RANDOMIZED, OPEN LABEL STUDY OF PROLONGED THERAPY WITH SC BORTEZOMIB TWICE MONTHLY ASSOCIATED WITH DEXAMETHASONE, IN RELAPSED AND REFRACTORY MULTIPLE MYELOMA PATIENTS AFTER SALVAGE WITH BORTEZOMIB-BASED THERAPY.
Brief Title: Maintenance Therapy With Subcutaneous Bortezomib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-MMY-2084
Record Dates: First submitted 2013-04-10; First posted 2013-08-01 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Refractory; Relapsed
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No prolonged therapy is scheduled (No Intervention)
- Bortezomib Dexamethasone (Biochemical relapse) (Experimental): Patients randomized in this group will be observed. At the occurrence of biochemical relapse, 4 VD cycles will be administered: Bortezomib (SC) and Dexamethasone (PO) weekly.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib
  Arms: Bortezomib Dexamethasone (Biochemical relapse)
Drug: Dexamethasone
  Arms: Bortezomib Dexamethasone (Biochemical relapse)

SUMMARY:
This is a multicenter, randomized, open label study designed to evaluate the efficacy and safety of prolonged treatment with bortezomib twice monthly and dexamethasone after a salvage treatment containing bortezomib for relapsed or refractory multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is of a legally consenting age as defined by local regulations.
2. Patient is, in the investigator(s) opinion willing and able to comply with the protocol requirements.
3. Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
4. Female patient is either post-menopausal for 24 consecutive months or surgically sterilised or agree to continuous abstinence from heterosexual sexual contact or willing to use two acceptable method of birth control at the same time (one highly effective method and one additional effective method) (Highly Effective Methods: Intrauterine device -IUD-; Hormonal -birth control pills, injections, implants-; tubal ligation; partner's vasectomy; Additional Effective Methods: Latex condom; Diaphragm; Cervical Cap) for 4 weeks prior to beginning study drug therapy, during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of therapy.
5. Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) during study drug therapy (including dose interruption) and for 4 weeks after discontinuation of bortezomib therapy.
6. Patient was previously diagnosed with multiple myeloma based on standard criteria.
7. Patient is relapsed or refractory after one to three lines of treatment and the last one must be a bortezomib-containing regimen, without evidence of progressive disease.
8. Patient had previously received at least 4 cycles of a salvage treatment containing bortezomib, before enrolment, without evidence of progressive disease.
9. Patient must be enrolled and start therapy within 45 days from the completion of the last salvage cycle containing Bortezomib.
10. Before the salvage treatment with bortezomib-based regimens, patient must have measurable disease

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality or psychiatric illness that prevented the subject from signing the informed consent form or placed the subjects at unacceptable risk.
2. Pregnant or lactating females
3. Known positive for HIV or active infectious hepatitis type A, B or C
4. Peripheral neuropathy or neuropathic pain grade 2 or higher, as defined by National Cancer Institute Common Toxicity Criteria (NCI CTC) 4.0
5. Infiltrative pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Time to Progression | 5 years

SECONDARY OUTCOMES:
Survival | 5 years
  Overall Survival Progression Free Survival
Response | 5 years
  Objective overall response rate (ORR)
Response | 5 years
  Duration of response
Response | 5 years
  Time to response
Response | 5 years
  Time to the next anti-myeloma therapy (TNT)
Response | 5 years
  TTP measured from the beginning of the salvage treatment
Response | 5 years
  Role of the type of salvage treatment
Response | 5 years
  Role of previous treatments
Response | 5 years
  Incidence of grade 3 and 4 hematological and non-hematological adverse events (AEs)
Response | 5 years
  Exploratory assessment on prognosis (ISS, age and FISH abnormalities)

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Crob, Rionero in Vulture, Potenza, Italy